CLINICAL TRIAL: NCT05431686
Title: Group Visits to Improve Technology Use, Glycemic Control, and Quality of Life in High Risk Children With Type 1 Diabetes
Brief Title: Group Visits for High Risk Type 1 Diabetes (T1D)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: American Diabetes Association (Other); DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00016268
Record Dates: First submitted 2022-03-18; First posted 2022-06-24 (Actual); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: The study will include the intervention group participating in the SMA visits (n=20)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMA visit intervention arm (Experimental): SMAs will occur once every 3 months, and consist of 4-6 underserved youth with T1D and their primary diabetes caregiver
  Interventions: Behavioral: SMA visits

INTERVENTIONS:
Behavioral: SMA visits — SMA visit once every 3 months over a 12 month period

SUMMARY:
The investigators propose to conduct a pilot prospective cohort study to assess the impact of shared medical appointments (SMA) visits in underserved youth with poorly controlled type 1 diabetes (T1D). The trial will employ an enrollment visit, SMA visits every 3 months over a 12 month study period, followed by a 6-month observational period to assess feasibility and acceptability of SMA and the impact on glycemic control, self-management skills, and health related quality of life.

DETAILED DESCRIPTION:
Dyads of youth with T1D aged 8-12 years and their primary diabetes caretakers identifying as non-Hispanic Black or Latinx will be recruited to participate in a pilot prospective cohort study exploring feasibility and acceptability of SMA and the impact on glycemic control, self-management skills, and health related quality of life. This trial will employ an enrollment visit, SMA visits every 3 months over a 12-month study period, and a follow-up 6-month observational period to continue to evaluate outcomes once patients return to routine individual follow up care. The study will include the intervention group participating in the SMA visits (n=20).

All staff participating in the SMA visit will receive comprehensive training on how to facilitate the SMA discussion sessions effectively. All topics that will be covered at each SMA visit will be reviewed by the study staff ahead of the visit. Potential participants will be screened for participation using our electronic medical records system and will be approached during routine clinical visits. After explaining all study procedures, informed consent using an IRB-approved consent form will be obtained for all participants. After obtaining consent, a blinded Dexcom G6 CGM will be placed on the participant. Participants will be instructed to wear the blinded CGM for 10 days in order to obtain baseline glycemic control data prior to starting the SMA visit intervention. At the completion of the 10 day wear period, participants will mail back the blinded CGM in a pre-addressed envelope so that the data can be assessed within 30 days of the wear time. Because SMA visits will be used in place of routine clinic visits and because participants will not require any additional in person study visits, the investigators anticipate significant interest in participation with minimal barriers. Secure REDCap surveys will be sent to participants via email 1 week before each follow-up visit. If the surveys have not been completed at the time of the visit the participant will be asked to complete the measures using an iPad or paper in clinic at the time of their visit. Youth who elected not to use a CGM for routine clinical care, will be asked to wear a blinded professional CGM for 10 days prior to each visit whenever possible.

SMA Structure: SMAs will consist of 4-6 underserved youth with T1D and their primary diabetes caregiver. All youth and caretakers will complete standard check-in procedures with the clinic medical staff, including routine clinical intake questionnaires, vital sign assessments and point-of-care fingerstick A1c measurements. Before each session, dyads will be invited to submit questions to the research team that will then be anonymously reviewed and discussed among the group during the SMA. In the event that no questions are submitted by families, the facilitator will begin the discussion with stories and questions related to technology use and potential barriers in order to focus the discussion on the aspect of diabetes management being highlighted in that specific SMA. After discussing the questions, the facilitator will lead a group discussion focusing on the topic of the day. During each visit, the facilitator role will be shared by a pediatric endocrinologist, CDCES, nutritionist, and psychologist. Youth and caregivers will individually meet with the endocrinologist at different time points during the session to update personal management plans and goals of care. The group visit will conclude with a review of the core concepts discussed. Youth will be encouraged to set and share individual goals to be addressed before the next SMA.

Enrollment visit: This visit will occur at a routine clinic visit once a patient expresses interest in participating in the study. Alternatively, patients expressing interest in enrolling who are unable to do so at a routine clinic visit will have the option to come back for enrollment at a different time. A study team member will meet with the patient and family to review the study details and obtain consent. A blinded Dexcom G6 pro CGM will be placed on the patient and be worn for 10 days in order to collect baseline data prior to starting the intervention. Phone applications that will allow for sharing of CGM data between patients and the diabetes clinical care team will be downloaded and established before the end of the visit.

Initial SMA: The structure of the group visits will be reviewed with patients and families, and all members of the diabetes team will introduce themselves and explain their role in diabetes care. As some patients will be CGM naïve before this visit, education will focus on insertion and removal of the CGM along with appropriate use of the CGM receiver, alerts and alarms, data sharing, and troubleshooting common CGM problems. Established sharing of CGM data between patients and the diabetes clinical care team will be confirmed before the end of the visit. The group visit will conclude with a review of the core concepts discussed, and patients will set goals for the next SMA.

Follow Up SMA: Follow up SMA will be scheduled 3, 6, 9, and 12 months from the initial group visit. CGM data from 14 days prior to each SMA will be reviewed by the endocrinologist ahead of the group visit. Discussions and education guided by the facilitators will focus on issues that have been described in the literature as potential barriers to CGM use and adherence. Recurrent alerts and alarms can result in alarm fatigue, and falsely low glucose readings and sensor or transmitter failures have been cited as reasons for discontinuing CGM use. The continuous nature of CGM data has been shown to place significant demands on patients and their families, and to create stress related to the constant need for diabetes-related attention. Follow up visits will focus on optimized use of CGM alarms and prevention of alarm fatigue. Psychologists and CDCES will discuss strategies to cope with the on-body presence and potential embarrassment resulting from CGM wear and to optimize parent-child communication surrounding CGM. Nutritionists will highlight the impact of different foods on glycemic trends and discuss strategies to optimize control. SMA will also allow ample opportunity to jointly review de-identified CGM reports and how to effectively interpret data and make management changes in response to CGM data, empowering patients and families to improve self-management and reduce stress related to CGM use. Active participation in discussions and group exercises will continue to strengthen the community feeling and social support network within the SMA group. Any participant that chooses to discontinue CGM during the 12 month study period will wear a blinded CGM 10 days prior to the follow up visits to allow for complete data collection. Upon completion of the final SMA visit at month 12, dyads will be contacted to schedule a semi-structured interview and will then return to standard clinical care.

3-Month and 6-Month Post-Intervention Follow-Ups: Survey measures and assessments of glycemic control will be repeated after 3 months and 6 months of routine clinical care to assess for long-lasting effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically diagnosed with T1D managed with insulin injections for at least 1 year
* Non-Hispanic Black or Latinx ethnicity
* Public healthcare insurance
* Male or female ages ≥ 8 and < 12 years
* Poorly controlled T1D: one A1c value > 8% in the preceding year
* Fluent in English as the Dexcom technology is currently available only in English
* Participation of the primary diabetes caregiver

Exclusion Criteria:

* Use of insulin pump therapy for diabetes management at time of enrollment
* Major illnesses other than T1D
* Significant cognitive limitations and major psychiatric disorders in the child or
* Concurrent use of any non-insulin diabetes medication to control blood glucose levels.
* Concurrent participation in any other clinical studies during study period

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shideh Majidi, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giani E, Snelgrove R, Volkening LK, Laffel LM. Continuous Glucose Monitoring (CGM) Adherence in Youth With Type 1 Diabetes: Associations With Biomedical and Psychosocial Variables. J Diabetes Sci Technol. 2017 May;11(3):476-483. doi: 10.1177/1932296816676280. Epub 2016 Nov 1. PMID 27807014
- [Background] Jeon, Jouhyun, et al.
- [Background] Hilliard ME, Levy W, Anderson BJ, Whitehouse AL, Commissariat PV, Harrington KR, Laffel LM, Miller KM, Van Name M, Tamborlane WV, DeSalvo DJ, DiMeglio LA. Benefits and Barriers of Continuous Glucose Monitoring in Young Children with Type 1 Diabetes. Diabetes Technol Ther. 2019 Sep;21(9):493-498. doi: 10.1089/dia.2019.0142. Epub 2019 Jul 9. PMID 31287721
- [Derived] Grundman JB, Majidi S, Perkins A, Streisand R, Monaghan M, Marks BE. Applying the use of shared medical appointments (SMAs) to improve continuous glucose monitor (CGM) use, glycemic control, and quality of life in marginalized youth with type 1 diabetes: Study protocol for a pilot prospective cohort study. Contemp Clin Trials Commun. 2023 Jan 16;32:101067. doi: 10.1016/j.conctc.2023.101067. eCollection 2023 Apr. PMID 36698741

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: all participants are assigned to a single SMA visit intervention arm
Period: Overall Study
Arm/Group | SMA Visit Intervention Arm
Started | 14 (14 youth, 14 caregivers)
Completed | 4 (4 youth, 4 caregivers)
Not Completed | 10
Not completed — unable to schedule | 10

BASELINE CHARACTERISTICS:
Population: baseline characteristics were collected from youth only, not from caregivers
Groups:
- SMA Visit Intervention Arm: SMAs will occur once every 3 months, and consist of 4-6 underserved youth with T1D and their primary diabetes caregiver. Baseline characteristic data was collected for youth, not from caregivers.
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eligible Participants Who Agreed to Participate as Assessed by Tracking Those Who Were Approached to Participate and Those Who Agreed to Participate
Description: Investigators will track all patients who screened eligible to participate in the study, as well as those who that were contacted to gauge interest in participating. Investigators will track the percent of people who agreed to participate from those that were approached, with the goal of >60% of those reached/eligible to participate agreeing to enroll as a measure of feasibility.
Time Frame: 12 months
Population: Inclusion criteria: ages 8-12 years, Non-Hispanic Black (NHB) or Latinx, publicly insured, insulin pump naïve, recent HbA1c >8%
Measure: Count of Participants; unit: Participants
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 82
Participants | 14

2. Primary Outcome: Percentage of Participants With CGM Use, as Assessed by Tracking CGM Use Status From Enrollment to the End of the Study.
Description: For those who agree to enroll, investigators will classify participant's CGM use status at time of enrollment as either current CGM users, never CGM users, or those with CGM attrition. At the completion of the study, CGM use status will be assessed, with the goal of >80% current CGM users among study participants as a measure of feasibility.
Time Frame: 18 months
Population: SMA intervention participants
Measure: Median (Inter-Quartile Range); unit: percentage of 14 day CGM wear
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 4
percentage of 14 day CGM wear | 87.5 [80.1 to 92.7]

3. Primary Outcome: Frequency of SMA Sessions Attended, as Assessed by Tracking Study Visit Attendance.
Description: For those who agree to enroll, investigators will document if participants attended or were absent from scheduled study visits. At the completion of the study, attendance will be assessed, with the goal of >80% sessions attended among study participants as a measure of feasibility.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: percentage of visits attended
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 4
percentage of visits attended | 90 [80 to 100]

4. Primary Outcome: Perceived Satisfaction of SMA Intervention as Assessed by Semi-structured Interviews.
Description: Thematic analysis of qualitative data will be conducted by two team members who independently review interview transcripts to generate initial codes. Initial codes will be discussed by the group to generate a list of second-cycle codes and each team member will then apply coding framework to all transcripts before identifying dominant themes. ATLAS.ti software will be used to organize and analyze qualitative data.
Time Frame: 12 months
Population: 2 youth-caregiver dyads participated in semi-structured interviews
Measure: Count of Participants; unit: Participants
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 2
Participants | 2

5. Primary Outcome: Perceived Utility of the SMA Intervention Content, as Measured by User Satisfaction Surveys Summary Statistics (Mean and Standard Deviation as Well as Percent Answering a Specific Likert Level)
Description: Youth and caregivers randomized to the SMA intervention will complete user satisfaction ratings at the end of the SMA intervention to evaluate intervention utility. Investigators will report results of the satisfaction ratings, with the goal of >80% reporting perceived utility as a measure of acceptability.
Time Frame: 12 months
Population: user satisfaction ratings were not collected given the small study sample population, instead, semi-structured interviews were performed to collect acceptability data
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 0

6. Primary Outcome: Perceived Benefit of the SMA Intervention Content, as Measured by User Satisfaction Surveys Summary Statistics (Mean and Standard Deviation as Well as Percent Answering a Specific Likert Level)
Description: Youth and caregivers randomized to the SMA intervention will complete user satisfaction ratings at the end of the SMA intervention to evaluate intervention benefit. Investigators will report results of the satisfaction ratings, with the goal of >80% reporting perceived benefit as a measure of acceptability.
Time Frame: 12 months
Population: as for outcome 5
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 0

7. Secondary Outcome: Percentage of Time in Range (70-180 mg/dl)
Description: We will look at differences in the percent of time that blood sugar values are in range within subject measures across the SMA intervention and during the follow up period.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
Population: given the small sample size, there is not sufficient power to evaluate changes over time so statistical analysis was not performed for this outcome
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 4
percentage of time
  Baseline | 27.25 (1.71)
  3 months | 21.75 (10.56)
  6 months | 23.67 (3.79)
  9 months | 29.00 (5.66)
  12 months | 33.33 (8.33)
  15 months | 38.00 (3.61)
  18 months | 27.00 (9.17)

8. Secondary Outcome: Continuous Glucose Monitor Time Below Range (<70 mg/dL)
Description: We will look at differences in the percent of time that blood sugar values are below range within subject measures across the SMA intervention and during the follow up period.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of time below range
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 4
percentage of time below range
  Baseline | 2.45 (1.73)
  3 months | 0.97 (1.00)
  6 months | 4.00 (4.58)
  9 months | 2.00 (0.00)
  12 months | 1.60 (1.47)
  15 months | 2.50 (0.71)
  18 months | 1.67 (2.08)

9. Secondary Outcome: Continuous Glucose Monitor Time Above Range (>180 mg/dL)
Description: We will look at differences in the percent of time that blood sugar values are above range within subject measures across the SMA intervention and during the follow up period.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of time above range
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 4
percentage of time above range
  baseline | 78.00 (15.62)
  3 months | 80.77 (10.51)
  6 months | 72.33 (8.33)
  9 months | 69.00 (5.66)
  12 months | 61.33 (20.03)
  15 months | 60.00 (4.24)
  18 months | 71.00 (11.53)

10. Secondary Outcome: Continuous Glucose Monitor Mean Sensor Glucose
Description: We will look at differences in the mean sensor glucose values within subject measures across the SMA intervention and during the follow up period.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 4
mg/dl
  baseline | 247.75 (17.75)
  3 months | 259.25 (35.51)
  6 months | 245.33 (13.05)
  9 months | 241.50 (3.54)
  12 months | 239.00 (30.51)
  15 months | 219.67 (15.82)
  18 months | 256.67 (47.51)

11. Secondary Outcome: Continuous Glucose Monitor Coefficient of Variation
Description: We will look at differences in the coefficient of variation values within subject measures across the SMA intervention and during the follow up period.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 4
percentage
  baseline | 41.40 (7.38)
  3 months | 30.80 (7.75)
  6 months | 41.47 (12.52)
  9 months | 42.30 (4.67)
  12 months | 43.30 (9.36)
  15 months | 44.85 (3.61)
  18 months | 39.40 (5.63)

12. Secondary Outcome: Continuous Glucose Monitor Wear Time
Description: We will look at differences in percent CGM wear time within subject measures across the SMA intervention and during the follow up period.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of CGM wear time
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 4
percentage of CGM wear time
  baseline | 63.40 (16.75)
  3 months | 67.33 (19.79)
  6 months | 64.33 (44.84)
  9 months | 89.50 (4.95)
  12 months | 74.00 (27.07)
  15 months | 71.13 (18.80)
  18 months | 65.90 (23.08)

13. Secondary Outcome: Episodes of Diabetic Ketoacidosis (DKA)
Description: We will look at differences in number of episodes of DKA since the last study visit within subject measures across the SMA intervention and during the follow up period.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: DKA episodes
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 4
DKA episodes
  baseline | 0 (0)
  3 months | 0 (0)
  6 months | 0 (0)
  9 months | 0 (0)
  12 months | 0 (0)
  15 months | 0 (0)
  18 months | 0 (0)

14. Secondary Outcome: Episodes of Severe Hypoglycemia
Description: We will look at differences in number of episodes of severe hypoglycemia since the last study visit within subject measures across the SMA intervention and during the follow up period.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: severe hypoglycemia episodes
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 4
severe hypoglycemia episodes
  baseline | 0 (0)
  3 months | 0 (0)
  6 months | 0 (0)
  9 months | 0 (0)
  12 months | 0 (0)
  15 months | 0 (0)
  18 months | 0 (0)

15. Secondary Outcome: Number of Emergency Room Visits
Description: We will look at differences in number of episodes of emergency room visits since the last study visit within subject measures across the SMA intervention and during the follow up period.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: emergency room visit episodes
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 4
emergency room visit episodes
  baseline | 0 (0)
  3 months | 0.5 (1.0)
  6 months | 0 (0)
  9 months | 0 (0)
  12 months | 0 (0)
  15 months | 0 (0)
  18 months | 0 (0)

16. Secondary Outcome: Number of Hospital Admissions
Description: We will look at differences in number of hospital admissions since the last study visit within subject measures across the SMA intervention and during the follow up period.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hospital admissions
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 4
hospital admissions
  baseline | 0 (0)
  3 months | 0 (0)
  6 months | 0 (0)
  9 months | 0 (0)
  12 months | 0 (0)
  15 months | 0 (0)
  18 months | 0 (0)

17. Secondary Outcome: Hemoglobin A1c
Description: We will look at differences in HbA1c at study visits within subject measures across the SMA intervention and during the follow up period.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | SMA Visit Intervention Arm
Number analyzed (Participants) | 4
percentage of HbA1c
  baseline | 11.28 (1.24)
  3 months | 10.60 (1.26)
  6 months | 10.47 (2.04)
  9 months | 9.35 (0.64)
  12 months | 9.67 (0.81)
  15 months | 10.70 (2.46)
  18 months | 10.70 (1.22)

18. Secondary Outcome: Type 1 Diabetes and Life (T1DAL) Survey
Description: The T1DAL is a validated survey assessing diabetes specific quality of life. Scores range from 0 to 100, with higher scores reflecting greater quality of life. Surveys will be completed at each of the study visits, and scores will be compared within subject measures across the SMA intervention and during the follow up period.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SMA Visit Intervention Arm - Youth; SMA Visit Intervention Arm - Caregiver: SMAs will occur once every 3 months, and consist of 4-6 underserved youth with T1D and their primary diabetes caregiver
  SMA visits: SMA visit once every 3 months over a 12 month period
Arm/Group | SMA Visit Intervention Arm - Youth | SMA Visit Intervention Arm - Caregiver
Number analyzed (Participants) | 4 | 4
score on a scale
  baseline | 67.95 (6.91) | 74.70 (11.39)
  3 months | 66.63 (10.44) | 72.32 (15.01)
  6 months | 68.45 (9.26) | 76.49 (16.65)
  9 months | 69.31 (5.04) | 75.40 (17.83)
  12 months | 63.51 (6.69) | 74.70 (15.01)
  15 months | 59.23 (9.93) | 77.78 (9.25)
  18 months | 62.82 (7.46) | 75.00 (17.47)

19. Secondary Outcome: Diabetes Self-Management Profile (DSMP) Survey
Description: The DSMP is a validated survey assessing T1D adherence. Scores range from 0 to 90, with higher scores reflecting better T1D management. Surveys will be completed at each of the study visits, and scores will be compared within subject measures across the SMA intervention and during the follow up period.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SMA Visit Intervention Arm - Youth | SMA Visit Intervention Arm - Caregiver
Number analyzed (Participants) | 4 | 4
score on a scale
  baseline | 47.97 (9.37) | 42.44 (10.42)
  3 months | 37.65 (7.3) | 65.41 (38.46)
  6 months | 33.58 (6.39) | 38.95 (27.66)
  9 months | 42.21 (11.32) | 42.64 (10.80)
  12 months | 40.03 (13.41) | 44.19 (10.70)
  15 months | 30.51 (7.46) | 37.98 (13.38)
  18 months | 38.23 (11.2) | 42.15 (9.37)

20. Secondary Outcome: Self-Efficacy for Diabetes Scale (SED) Survey
Description: The SED is a validated survey assessing diabetes-specific self-efficacy. Scores range from 0-4 for each question, with higher scores indicating increasing levels of child responsibility. The total scores can range from 0-100. Surveys will be completed at each of the study visits, and scores will be compared within subject measures across the SMA intervention and during the follow up period.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SMA Visit Intervention Arm - Youth | SMA Visit Intervention Arm - Caregiver
Number analyzed (Participants) | 4 | 4
score on a scale
  baseline | 45.84 (12.64) | 70.23 (7.17)
  3 months | 65.29 (4.9) | 68.41 (9.22)
  6 months | 53.77 (27.08) | 65.91 (10.64)
  9 months | 57.21 (18.87) | 63.94 (14.09)
  12 months | 70.6 (7.68) | 69.32 (9.91)
  15 months | 73.17 (8.74) | 72.12 (9.33)
  18 months | 68.12 (14.19) | 67.05 (9.01)

21. Secondary Outcome: Problem Areas in Diabetes (PAID) Scale
Description: The Problem Areas in Diabetes (PAID) scale is widely used for measuring diabetes-related emotional distress. Scores range from 0-5 for each question, with higher scores indicating greater burden relating to having diabetes. The total scores can range from 0-80. Surveys will be completed at each of the study visits, and scores will be compared within subject measures across the SMA intervention and during the follow up period.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SMA Visit Intervention Arm - Youth | SMA Visit Intervention Arm - Caregiver
Number analyzed (Participants) | 4 | 4
score on a scale
  baseline | 50.0 (16.96) | 59.69 (10.38)
  3 months | 50.66 (21.8) | 64.06 (10.48)
  6 months | 27.28 (36.0) | 67.81 (18.72)
  9 months | 44.09 (28.07) | 60.83 (6.41)
  12 months | 48.18 (25.74) | 64.06 (16.88)
  15 months | 49.04 (22.64) | 65.00 (13.75)
  18 months | 47.88 (14.58) | 61.25 (4.79)

22. Secondary Outcome: CGM Benefits and Burdens Scale
Description: The CGM Benefits and Burdens scale is widely used for measuring perceptions of CGM benefit and burdens. Raw scores range from 1-5 for each question, with higher scores reflecting greater burdens/benefits. Total scores are scaled and combined, ranging from 0-200. Surveys will be completed at each of the study visits, and scores will be compared within subject measures across the SMA intervention and during the follow up period.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SMA Visit Intervention Arm - Youth | SMA Visit Intervention Arm - Caregiver
Number analyzed (Participants) | 4 | 4
score on a scale
  baseline | 133.12 (48.5) | 81.25 (31.19)
  3 months | 96.25 (23.56) | 68.13 (32.87)
  6 months | 108.12 (2.65) | 46.88 (37.99)
  9 months | 103.44 (18.21) | 62.50 (26.34)
  12 months | 100.0 (16.36) | 54.38 (15.19)
  15 months | 87.5 (7.5) | 39.17 (1.44)
  18 months | 97.5 (15.21) | 51.88 (22.30)

ADVERSE EVENTS:
Time Frame: from enrollment until the end of follow up, up to 18 months
Groups:
- SMA Visit Intervention Arm - Youth; SMA Visit Intervention Arm - Caregivers: SMAs will occur once every 3 months, and consist of 4-6 underserved youth with T1D and their primary diabetes caregiver
Arm/Group | SMA Visit Intervention Arm - Youth | SMA Visit Intervention Arm - Caregivers
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
limited sample size as enrollment was challenging and there was a limited subset of participants who completed the protocol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT05431686/Prot_SAP_003.pdf